CLINICAL TRIAL: NCT01089296
Title: Parental Participation in Individually Customized Physiotherapy for Preterm Infants in the Neonatal Intensive Care Unit: Effects and Experiences. The Pragmatic Randomized Controlled Part.
Brief Title: The Norwegian Physical Therapy Study in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); St. Olavs Hospital (Other); University of Illinois at Chicago (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/370-00/09-A
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2021-03

CONDITIONS: Movement Disorders
Keywords: Infants born preterm; Early physiotherapy intervention; Motor development; Parental participation; Parental competency
MeSH Terms: conditions — Movement Disorders | interventions — Physical Therapy Modalities; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individually customized physiotherapy (Other): The intervention involves handling the infant and changing its position. It focuses on improving symmetry, muscle balance and movement in infants. The parent who is with the infant during the admission period will carry out the daily intervention after being taught by the physiotherapist.
  Interventions: Other: Individually customized physiotherapy
- Control (No Intervention): Ordinary follow up in the Neonatal Intensive Care Unit (NICU).

INTERVENTIONS:
Other: Individually customized physiotherapy — Main elements in the intervention are postural support and facilitating techniques. The intervention will be carried out twice a day over a three-week period if the infant's condition allows it. The length of each treatment session will be adjusted dependent on the infant's response and condition. Maximum treatment time is 10 minutes.
  Other Names: Physiotherapy; Physical Therapy; Premature birth; Early Intervention
  Arms: Individually customized physiotherapy

SUMMARY:
This is a pragmatic randomized controlled study. The purpose of the study is to evaluate the practice and effect of customised physiotherapy on preterm infants'motor development when the intervention is performed over a period of three weeks while the infant resides in the neonatal intensive care unit. The study will also attempt to analyze the parents' experiences in being actively involved in education and practice of the intervention designed to promote the child's motor development, and the effects on the parent-child relationship in the short and long term.The children are followed up until a corrected age of two years. This study consists of a pragmatic randomized controlled trial and a qualitative study.

DETAILED DESCRIPTION:
Infants born preterm with an gestational age below 32 weeks have an increased risk of developing different grades and types of abnormalities, among them delayed motor development, co-ordination difficulties and cerebral palsy. The prevalence of serious developmental abnormalities increases the lower the gestational age and birth weight. The reported incidence of mild developmental abnormalities is 15-20 % in children with a gestational age <28 weeks or with a birth weight under 1000 g, 10-20 % in children with a gestational age of 28-31 weeks or a birth weight between 1000-1500 g and only 5 % in children born at term. The incidence of cerebral palsy is 10-20% amongst children in the first group, 5-10% in the second group and only 0,1 % in children born at term.With such a high risk of developing motor abnormalities for infants born preterm together with limited evidence-based knowledge of early physiotherapy approaches that facilitate motor development, it is essential that more research is done in this area to ensure that physiotherapy if used, is in the right manner to prevent and reduce such difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Child born before or at 32nd gestational week.
* Child that tolerates being handled at 34th week postmenstrual age.
* Parents that can perform the intervention understand and speak Norwegian.
* Follow up of the child in the hospital where the intervention is given.

Exclusion Criteria:

* Child born later than 32nd week.
* Child who cannot tolerate being handled for up to 10 minutes at 34th postmenstrual age.
* Triplets or more.
* Child who has undergone surgery.
* Child with large deformities.
* Parents that can perform the intervention but do not understand and speak Norwegian.
* Follow up of the child is not taking place in the hospital where the intervention is given.
* All children who fill the inclusion criteria will be included to begin with.
* If at a later stage they are unable to manage the tests due to their condition they will be excluded.

Ages: 7 Days to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2010-03-18 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales(PDMS-2) | Two years post term age
  PDMS-2 assess both fine- and gross motor function. Even though our Primary Outcome Measure is at two years post term age, we are going to publish results from assessments at earlier ages when they exist for the whole sample as the study proceeds.

SECONDARY OUTCOMES:
Test of Infant Motor Performance Screening Items (TIMPSI), General Movement Assessment (GMA),Test of Infant Motor Performance(TIMP), Alberta Infant Motor Scale (AIMS), Peabody Developmental Motor Scales (PDMS-2) | TIMPSI: 34 w (baseline). GMA: 34 w, 36 w, 3 mo. TIMP: 37 w, 3 mo. AIMS: 3 mo, 6 mo, 12 mo. PDMS-2: 6 mo, 12 mo, 24 mo.
  Results from the different Time Frames will be published successively as the project proceeds.

CONTACTS AND LOCATIONS:
Overall Officials: Gunn K. Øberg, PhD, Principal Investigator — University of Tromsø / University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

REFERENCES:
- [Derived] Orton J, Doyle LW, Tripathi T, Boyd R, Anderson PJ, Spittle A. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2024 Feb 13;2(2):CD005495. doi: 10.1002/14651858.CD005495.pub5. PMID 38348930
- [Derived] Ustad T, Brandal M, Campbell SK, Girolami GL, Sinding-Larsen C, Oberg GK. Concurrent and predictive validity of the Alberta Infant Motor Scale and the Peabody Developmental Motor Scales-2 administered to infants born preterm in Norway. BMC Pediatr. 2023 Nov 23;23(1):591. doi: 10.1186/s12887-023-04402-6. PMID 37993837
- [Derived] Oberg GK, Girolami GL, Campbell SK, Ustad T, Heuch I, Jacobsen BK, Kaaresen PI, Aulie VS, Jorgensen L. Effects of a Parent-Administered Exercise Program in the Neonatal Intensive Care Unit: Dose Does Matter-A Randomized Controlled Trial. Phys Ther. 2020 May 18;100(5):860-869. doi: 10.1093/ptj/pzaa014. PMID 31944250
- [Derived] Ustad T, Evensen KA, Campbell SK, Girolami GL, Helbostad J, Jorgensen L, Kaaresen PI, Oberg GK. Early Parent-Administered Physical Therapy for Preterm Infants: A Randomized Controlled Trial. Pediatrics. 2016 Aug;138(2):e20160271. doi: 10.1542/peds.2016-0271. PMID 27440658
- [Derived] Oberg GK, Campbell SK, Girolami GL, Ustad T, Jorgensen L, Kaaresen PI. Study protocol: an early intervention program to improve motor outcome in preterm infants: a randomized controlled trial and a qualitative study of physiotherapy performance and parental experiences. BMC Pediatr. 2012 Feb 15;12:15. doi: 10.1186/1471-2431-12-15. PMID 22336194